CLINICAL TRIAL: NCT01357577
Title: CBT for PTSD in Veterans With Co-Occurring Substance Use Disorders
Brief Title: Cognitive Behavioral Therapy (CBT) for PTSD in Veterans With Co-Occurring SUDs
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLA-01-S09
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: PTSD; Substance Use Disorders
Keywords: PTSD; Substance Use Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: TAU + CBT (Experimental): The experimental group will receive treatment as usual (TAU) plus cognitive behavioral therapy (CBT).
  Interventions: Behavioral: Cognitive behavioral therapy for PTSD
- Arm 2: TAU (No Intervention): The "no intervention" group will receive treatment as usual (TAU).

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for PTSD — The CBT for PTSD model is based on modern theories of posttraumatic reactions that place a premium on the importance of individuals' appraisals of traumatic events, their own reactions and those of others, and the meaning of the experience in terms of oneself and one's place in the world. In addition, the model employs cognitive restructuring to teach individuals how to examine and challenge their trauma-related appraisals.
  Arms: Arm 1: TAU + CBT

SUMMARY:
With this research, the investigators hope to learn if cognitive behavioral therapy (CBT) for posttraumatic stress disorder (PTSD) works in people who have both PTSD and problems with drugs or alcohol. In the past, people who had problems with drugs and alcohol were not given treatment for their PTSD. It was believed that PTSD treatment would get in the way of their drug and alcohol treatment. Now the investigators believe that the PTSD symptoms may make it harder to avoid using drugs and alcohol, so the investigators want to see if people can get treatment for both problems at the same time.

One hundred-sixty Veterans from 3 sites who have both PTSD and substance use disorders will be in the study. In order to know if the PTSD treatment is helpful, half of the Veterans in this study will receive PTSD treatment and half will continue to get their usual mental health and/or substance abuse treatment. Who gets which treatment will be decided by a random process. The investigators will then compare the 2 groups to see if there are differences in their PTSD symptoms.

DETAILED DESCRIPTION:
A randomized clinical trial to evaluate the effectiveness of a relatively simple, manual-guided cognitive behavioral therapy (CBT) for PTSD in patients with substance use disorders (SUDs). One hundred sixty outpatients with comorbid PTSD and SUDs from three VA facilities will be randomly assigned to receive either CBT for PTSD in conjunction with standard treatment as usual (TAU) (n = 80) or TAU only (n = 80).

ELIGIBILITY:
Inclusion Criteria:

* At least age 18.
* Current SUD diagnosis.
* Score of at least 45 on CAPS.
* Must speak English.
* Must agree to be taped.

Exclusion Criteria:

* Acute psychotic symptoms, if not well connected with appropriate mental health services.
* Severe suicidality.
* Individuals with unstable medical or legal situations that would make completion of the study highly unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Hamblen, PhD, Principal Investigator — White River Junction VA Medical Center, White River Junction, VT
Locations (3):
- United States (3):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three Veteran Affairs Medical Centers (VAMC): Syracuse, NY VAMC; Tampa Bay, FL VAMC; and White River Junction, VT VAMC. Participants were recruited from outpatient and inpatient clinics at the three respective facilities.
Groups:
- Cognitive Behavioral Therapy (CBT) + Treatment as Usual (TAU): The experimental group will receive treatment as usual (TAU) plus cognitive behavioral therapy (CBT).
  Cognitive behavioral therapy for PTSD: The CBT for PTSD model is based on modern theories of posttraumatic reactions that place a premium on the importance of individuals' appraisals of traumatic events, their own reactions and those of others, and the meaning of the experience in terms of oneself and one's place in the world. In addition, the model employs cognitive restructuring to teach individuals how to examine and challenge their trauma-related appraisals.
- Treatment as Usual (TAU): The "no intervention" group will receive treatment as usual (TAU).
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) + Treatment as Usual (TAU) | Treatment as Usual (TAU)
Started | 64 | 65
Post-Treatment Assessment Completed | 24 | 39
Completed (Completed Milestone is defined at 6-month assessment completed) | 27 | 39
Not Completed | 37 | 26
Not completed — Lost to Follow-up | 20 | 16
Not completed — Withdrawal by Subject | 16 | 8
Not completed — look at data in database? | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Behavioral Therapy + Treatment as Usual: The experimental group will receive treatment as usual (TAU) plus cognitive behavioral therapy (CBT).
  Cognitive behavioral therapy for PTSD: The CBT for PTSD model is based on modern theories of posttraumatic reactions that place a premium on the importance of individuals' appraisals of traumatic events, their own reactions and those of others, and the meaning of the experience in terms of oneself and one's place in the world. In addition, the model employs cognitive restructuring to teach individuals how to examine and challenge their trauma-related appraisals.
- Treatment as Usual: The "no intervention" group will receive treatment as usual (TAU) without additional individual treatment..
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy + Treatment as Usual | Treatment as Usual | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 65 | 129
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age (years) | 42.2 (12.5) | 45.9 (11.5) | 44.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 61 | 61 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 57 | 58 | 115
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 19 | 34
  White | 46 | 42 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants] — As previously indicated, all participants were recruited three VAMCs in the United States: Syracuse, NY; White River Junction, VT; and Tampa, FL.
  Participants
    United States | 64 | 65 | 129

OUTCOME MEASURES:

1. Primary Outcome: CAPS Total Score Analysis Among Participants Completing at Least One Follow-up Assessment.
Description: PTSD symptom severity will be measured by the Clinician Administered PTSD Scale (CAPS). The Clinician Administered PTSD SCALE (CAPS) is the gold standard in PTSD assessment. It is a structured interview that can be used to: Make current (past month) diagnosis of PTSD and Make lifetime diagnosis of PTSD. The minimum value is a 0 and the maximum is 135, the higher the score the worse the outcome, i.e. the more severe PTSD.
Time Frame: Conclusion of treatment (post-treatment occurs approximately 4-months after treatment conclusion) and 6 months follow-up
Population: Our intention-to-treat analysis has N=80 patients (33 CBT; 47 control): It consists of patients with at least one follow-up (post or 6-mo) assessment (e.g., of the 64 participants randomized to CBT, 24 and 27 had a CAPS assessment at post and 6 months, respectively, with 33 participants having at least one valid follow-up CAPS).
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Treatment as Usual: The "no intervention" group will receive treatment as usual (TAU) without additional treatment.
Arm/Group | Cognitive Behavioral Therapy + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 33 | 47
score on scale
  CAPS Total Baseline | 77.2 (18.4) | 78.0 (16.2)
  CAPS Total Post-Treatment: number analyzed (Participants) | 24 | 38
  CAPS Total Post-Treatment | 67.5 (26.3) | 71.0 (26.4)
  CAPS Total 6 Months: number analyzed (Participants) | 27 | 37
  CAPS Total 6 Months | 72.2 (21.6) | 62.9 (21.9)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .48, Mixed Models Analysis — P-Value show above is for post-assessment time point; Mixed-model p-values are adjusted for study site and the baseline total CAPS score
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .12, Mixed Models Analysis — The p-value shown above is for the 6-month time point; Mixed-model p-values are adjusted for study site and the baseline total CAPS score
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .65, Mixed Models Analysis — The p-value shown above refers to the treatment main effect
Statistical Analysis 4: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .072, Mixed Models Analysis — The p-value shown above refers to the timepoint main effect
Statistical Analysis 5: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .0050, Mixed Models Analysis; The p-value shown above refers to the interaction
Statistical Analysis 6: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .12, Mixed Models Analysis; The p-value shown above refers to the site main effect

2. Secondary Outcome: Addiction Severity Index (Alcohol Addiction)
Description: The ASI is a standardized, structured interview that assesses past 30 days problem severity in seven areas. These seven areas include medical, employment, drug, alcohol, legal, family/social and psychiatric status. Problem severity is rated on a scale of 0.0 - 1.0 with a higher score indicative of more problem severity. All scales have a range from 0 to 1.0.
Time Frame: Baseline, Post-Treatment (approximately 4-months after treatment conclusion), and 6-Months
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cognitive Behavioral Therapy + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 31 | 41
score on scale
  Alcohol Baseline | .25 (.22) | .25 (.25)
  Alcohol Post-Treatment | .13 (.17) | .17 (.22)
  Alcohol 6-Months | .18 (.18) | .20 (.27)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other — mixed-effects linear regression model adjusted for study site and the baseline value of the dependent variable; p = .12, Mixed Models Analysis — Post-treatment P-value; Mixed-model p-values are adjusted for study site and baseline ASI (Alcohol Use) score
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .84, Mixed Models Analysis — 6-month P-Value; Mixed-model p-values adjusted for study site and Baseline ASI (Alcohol Use) score
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .26, Mixed Models Analysis — treatment main effect; Mixed-model p-values adjusted for study site and Baseline ASI (Alcohol Use) score
Statistical Analysis 4: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .14, Mixed Models Analysis — Timepoint main effect P-value; Mixed-model p-values adjusted for study site and Baseline ASI (Alcohol Use) score
Statistical Analysis 5: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .29, Mixed Models Analysis — interaction; Mixed-model p-values adjusted for study site and Baseline ASI (Alcohol Use) score
Statistical Analysis 6: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .16, Mixed Models Analysis — Site main effect P-Value; Mixed-model p-values adjusted for study site and Baseline ASI (Alcohol Use) score

3. Secondary Outcome: Addiction Severity Index (Drug Use)
Description: as for outcome 2
Time Frame: Baseline, Post-Treatment (approximately 4-months after treatment conclusion), and 6-Months
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cognitive Behavioral Therapy + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 32 | 42
score on scale
  Drug Use Baseline | .17 (.18) | .10 (.11)
  Drug Use Post-Treatment | .09 (.18) | .08 (.13)
  Drug Use 6-Months | .11 (.15) | .04 (.08)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .66, Mixed Models Analysis — Post-treatment p-value; Mixed-model p-values are adjusted for study site and baseline ASI (drug score)
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .53, Mixed Models Analysis — 6-month P-Value; Mixed model p-values are adjusted for study site and baseline ASI (Drug Use) score
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .86, Mixed Models Analysis — Treatment main effect P-Value; Mixed model p-values are adjusted for study site and baseline ASI (Drug Use) score
Statistical Analysis 4: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .16, Mixed Models Analysis — Timepoint main effect P-Value; Mixed model p-values are adjusted for study site and baseline ASI (Drug Use) score
Statistical Analysis 5: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .47, Mixed Models Analysis — Interaction P-Value; Mixed model p-values are adjusted for study site and baseline ASI (Drug Use) score
Statistical Analysis 6: Comparison: Cognitive Behavioral Therapy + Treatment as Usual; Test type: Other; p = .19, Mixed Models Analysis — Site main effect P-Value; Mixed model p-values are adjusted for study site and baseline ASI (Drug Use) score

4. Secondary Outcome: PTSD Checklist (PCL)
Description: A secondary measure of PTSD will be the PCL. The PCL is a widely used self-report measure that assesses the 17 DSM-IV PTSD symptoms. Responses to these questions are on a scale of 1 to 5 ("not at all" to "extremely"). A total symptom severity score (range from 17-85) can be calculated, with a higher score indicating higher symptom severity.
Time Frame: Baseline, Post-Treatment (approximately 4-months post treatment completion), 6-months
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cognitive Behavioral Therapy + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 31 | 45
score on scale
  PCL Baseline | 62.7 (9.2) | 62.1 (13.3)
  PCL Post-Treatment | 54.3 (17.7) | 56.9 (15.7)
  PCL 6-months | 56.7 (13.7) | 54.2 (16.9)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .18, Mixed Models Analysis — Post-Treatment P-Value; Mixed model p-values are adjusted for study site and baseline PCL score
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .45, Mixed Models Analysis — P-value at 6 months; Mixed model p-values are adjusted for study site and baseline PCL score
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy + Treatment as Usual; Test type: Other; p = .73, Mixed Models Analysis — Treatment main effect P-Value; Mixed model p-values are adjusted for study site and baseline PCL score
Statistical Analysis 4: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .63, Mixed Models Analysis — Timepoint main effect P-Value; Mixed model p-values are adjusted for study site and baseline PCL score
Statistical Analysis 5: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .024, Mixed Models Analysis — Interaction P-Value; Mixed model p-values are adjusted for study site and baseline PCL score
Statistical Analysis 6: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .15, Mixed Models Analysis — Site main effect P-Value; Mixed model p-values are adjusted for study site and baseline PCL score

5. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: Patient Health Questionnaire-9 (PHQ-9): The PHQ-9 is adapted from the PRIME-MD. It can be used as a screen for depression or as a severity measure. The investigators used it as a measure of severity. The PHQ-9 score is on a range of 0 to 27, where a higher score indicates higher severity.
Time Frame: Baseline, Post-Treatment (approximately 4-months post treatment completion), 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy + Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 31 | 45
score on a scale
  PHQ-9 Baseline | 16.0 (4.7) | 14.8 (6.8)
  PHQ-9 Post-Treatment | 15.0 (7.4) | 12.8 (7.2)
  PHQ-9 6-months | 15.8 (17.1) | 12.2 (7.4)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .48, Mixed Models Analysis — Post-Treatment P-Value; Mixed model p-values are adjusted for study site and baseline PHQ score
Statistical Analysis 2: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .20, Mixed Models Analysis — 6-Month P-Value; Mixed model p-values are adjusted for study site and baseline PHQ score
Statistical Analysis 3: Comparison: Cognitive Behavioral Therapy + Treatment as Usual; Test type: Other; p = .26, Mixed Models Analysis — Treatment main effect P-Value; Mixed model p-values are adjusted for study site and baseline PHQ score
Statistical Analysis 4: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .71, Mixed Models Analysis — Timepoint main effect; Mixed model p-values are adjusted for study site and baseline PHQ score
Statistical Analysis 5: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .56, Mixed Models Analysis — Interaction main effect P-Value; Mixed model p-values are adjusted for study site and baseline PHQ score
Statistical Analysis 6: Comparison: Cognitive Behavioral Therapy + Treatment as Usual vs Treatment as Usual; Test type: Other; p = .51, Mixed Models Analysis — Site main effect P-Value; Mixed model p-values are adjusted for study site and baseline PHQ score

ADVERSE EVENTS:
Time Frame: Participants were monitored for both adverse events and serious adverse events (AE/SAE) once they were enrolled in the clinical trial. Assessors and clinical staff asked participants about any possible AE/SAE at post-assessment and 6-months. CBT+TAU clinical staff also asked participants about any AE/SAEs during their clinical sessions.
Description: Serious Adverse Events (SAEs) and Adverse Events (AEs) follow the definitions as outlined by clinicaltrials.gov but also VHA Handbook 1200.5:
Arm/Group | Cognitive Behavioral Therapy (CBT) + Treatment as Usual (TAU) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/64 | 1/65
Serious Adverse Events (participants affected / at risk) | 11/64 | 13/65
Other Adverse Events (participants affected / at risk) | 21/64 | 21/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (CBT) + Treatment as Usual (TAU) (N=64) | Treatment as Usual (TAU) (N=65)
Mental Health Episode resulting in hospital encounter (Psychiatric disorders) | 9 (9) | 7 (7)
Hospitalization for kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Hospitalization due to hip replacement surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
incarceration (Social circumstances) | 0 (0) | 1 (1)
inpatient stay for untreated COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Testicular and groin surgery resulting in inpatient hospital stay (Renal and urinary disorders) | 1 (1) | 0 (0)
hospitalization due to syncopal episode (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cognitive Behavioral Therapy (CBT) + Treatment as Usual (TAU) (N=64) | Treatment as Usual (TAU) (N=65)
Mental Health and/or Substance Abuse ER visit (Psychiatric disorders) | 10/10 (10) | 8 (8)
Jail (Social circumstances) | 1 (1) | 1 (1)
corneal abrasion (Eye disorders) | 1 (1) | 0 (0)
ER visit due to dental pain and/or possible dental abscess (General disorders) | 1 (1) | 1 (1)
chronic pain (General disorders) | 3 (3) | 1 (1)
musculature pain and discomfort (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
chest pain (Cardiac disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 2 (2)
hemophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
testicular pain (General disorders) | 0 (0) | 1 (1)
motor vehicle accident which results in paralysis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT01357577/Prot_SAP_000.pdf